CLINICAL TRIAL: NCT05399329
Title: Retrospective, Multicenter, Observational Study to Evaluate Real-World Effectiveness of Palbociclib Plus Endocrine Therapy in Japanese Patients With HR+/HER2- Advanced Breast Cancer in First Line or Second Line Settings
Brief Title: Study to Evaluate Real-world Effectiveness With Palbociclib Plus Endocrine Therapy as First-line/Second-line Treatment for HR+/HER2- Advanced Breast Cancer in Japan
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481166; NCT05399329 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Retrospective; Multicenter; Observational; Effectiveness; Real-world progression free survival; Palbociclib; Endocrine therapy; Japan; Hormone receptor positive/ human epidermal growth factor negative (HR+/HER2-); Advanced Breast Cancer; First-line therapy; Second-Line therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Palbociclib — Palbociclib plus ET as first-line/second-line treatment for hormone receptor positive/human epidermal growth factor receptor 2 negative (HR+/HER2-) ABC
Drug: Endocrine therapy — Palbociclib plus ET as first-line/second-line treatment for HR+/HER2- ABC

SUMMARY:
This is a retrospective, multicenter, observational study in Japan by medical record review of advanced breast cancer (ABC) patients who have received palbociclib plus endocrine therapy (ET) as first line or second line setting. For the purposes of this study, analyses will be descriptive in nature. No formal hypothesis testing is planned.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HR+/HER2- ABC
* Age of 20 years or older at diagnosis of ABC
* Patients that received palbociclib plus ET in the first line or second line
* Patients who meet the criteria regarding the medical record below:
* Patients with any medical records (regardless of palbociclib use) for more than 6 months from palbociclib initiation OR
* Patients with any medical records for less than 6 months from palbociclib initiation AND who had specific events (death, disease progression, or treatment discontinuation of palbociclib due to adverse events) in the available records

Exclusion Criteria:

* Patients who received chemotherapy as first line treatment.
* Patients who have previously participated or are participating in any interventional clinical trials that include investigational or marketed products.

(Interventional clinical trials for early breast cancer and later line after palbociclib will be acceptable, Besides, patients participating in other investigator-initiated research or noninterventional studies can be included as long as their standard of care is not altered by the study.)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study uses secondary data of multiple sites by utilizing medical record review approach for those who have been diagnosed with ABC in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 688 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Real-World Progression-Free Survival (rwPFS) of palbociclib plus ET as first line treatment for HR+/HER2- ABC | 15 December 2017 to 31 August 2023
rePFS of palbociclib plus ET as second line treatment for HR+/HER2- ABC | 15 December 2017 to 31 August 2023

SECONDARY OUTCOMES:
Landmark overall survival (OS) (defined from palbociclib initiation to death) of palbociclib plus ET as first line treatment for HR+/HER2- ABC | 15 December 2017 to 31 August 2023
Landmark OS (defined from palbociclib initiation to death)of palbociclib plus ET as second line treatment for HR+/HER2- ABC | 15 December 2017 to 31 August 2023
Landmark OS (defined from treatment initiation of first line to death) when palbociclib plus ET were used as second line treatment for HR+/HER2- ABC | 15 December 2017 to 31 August 2023
Time to treatment discontinuation (TTD) of palbociclib plus ET as first line or second line treatment for HR+/HER2- ABC | 15 December 2017 to 31 August 2023
TTD of first subsequent treatment for HR+/HER2- ABC patients who were treated with palbociclib plus ET | 15 December 2017 to 31 August 2023
Time to chemotherapy (TTC: defined as the time from treatment initiation of first or second line for HR+/HER2- ABC to first use of chemotherapy) | 15 December 2017 to 31 August 2023
Real-world objective response rate (rwORR) of palbociclib plus ET as first line or second line treatment for HR+/HER2- ABC | 15 December 2017 to 31 August 2023
Demographic of HR+/HER2- ABC patients who were treated with palbociclib plus ET in routine clinical practice in Japan | 15 December 2017 to 31 August 2023
Clinical characteristics of HR+/HER2- ABC patients who were treated with palbociclib plus ET in routine clinical practice in Japan | 15 December 2017 to 31 August 2023
Treatment patterns of palbociclib plus ET in routine clinical practice in Japan | 15 December 2017 to 31 August 2023

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- Japan (20):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Japan Community Health care Organization Kurume General Hospital, Kurume, Fukuoka
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Kaizuka City Hospital, Kaizuka, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Saitama Prefectural Cancer Center, Kita-adachi-gun, Saitama
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Gifu University Hospital, Gifu
  - Hiroshima University Hospital, Hiroshima
  - Tokai University Hospital, Kanagawa
  - Aichi Cancer Center, Nagoya
  - National Hospital Organization Osaka National Hospital, Osaka
  - Shizuoka Prefectural Hospital Organization, Shizuoka
  - Showa University Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481166